CLINICAL TRIAL: NCT05921162
Title: A Long-Term Follow-Up Study in Subjects Who Received an Adeno-Associated Viral Vector Serotype 2 Containing the Multi-Characteristic Opsin Gene (vMCO-I) Administered Via Intravitreal Injection
Brief Title: A Long-Term Follow-Up Study in Subjects Who Received vMCO-I Administered Via Intravitreal Injection
Acronym: EXTEND
Status: Enrolling by invitation | Type: Observational
Sponsor: Nanoscope Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NTXMCO-005
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Retinitis Pigmentosa; Retinal Disease; Retinal Degeneration
Keywords: Optogenetics; Gene Therapy; AAV Vectors; Multicharacteristic Opsin (MCO)-I
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; Retinal Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation of Participants exposed to 1.2E11gc/eye of vMCO-I: This is a long-term follow-up observational study of participants who previously received 1.2E11gc/eye of vMCO-I No investigational product will be administered in this study.
  Interventions: Biological: Gene Therapy product:vMCO-I
- Observation of Participants exposed to 0.6E11gc/eye of vMCO-I: This is a long-term follow-up observational study of participants who previously received 0.6E11gc/eye of vMCO-I No investigational product will be administered in this study.
  Interventions: Biological: Gene Therapy product:vMCO-I

INTERVENTIONS:
Biological: Gene Therapy product:vMCO-I — Safety evaluation to monitor long term effects of previously injected vMCO-I in RP patients

SUMMARY:
This study "A Long-Term Follow-Up Study in Subjects Who Received an Adeno-Associated Viral Vector Serotype 2 Containing the Multi-Characteristic Opsin Gene (vMCO-I) Administered Via Intravitreal Injection" is an observational study and will be conducted following Good Clinical Practice (GCP)- International Conference on Harmonization (ICH) guidelines. Eligible subjects satisfying all inclusion and none of the exclusion criteria will be enrolled. All subject who completed the parent clinical study (NSCT/CT/18/01) will undergo safety and efficacy assessments up to 5 years post study drug injection

DETAILED DESCRIPTION:
The observational study population comprises of individuals who received an Adeno-Associated Viral Vector Serotype 2 Containing the Multi-Characteristic Opsin Gene (vMCO-I) Administered Via Intravitreal Injection in a parent study.

Enrolled subjects will undergo safety and efficacy assessments for up to 5 years from the vMCO-I administration. At the visits, subjects will have safety and efficacy evaluations. Subjects will have a final visit at 60 months post study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* The subject population includes subjects who received an Adeno-Associated Viral Vector Serotype 2 Containing the Multi-Characteristic Opsin Gene (vMCO-I), administered via intravitreal injection in a parent study.

Exclusion Criteria:

* Subjects who will not consent for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is expected that a total of 11 study subjects from NSCT/CT/18/01 study will be enrolled. Subjects who meet all the inclusion criteria and for whom none of the exclusion criteria apply will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the long-term safety profile of a single intravitreal injection of vMCO-I | 20 Months
  Assessments of Incidences, nature, and severity of treatment emergent adverse events (TEAEs), Serious Adverse Events (SAEs); intraocular inflammation graded through ocular exam; intraocular pressure and retinal anatomy
Evaluation of the long-term efficacy of a single intravitreal injection of Multi-Characteristic Opsin (vMCO-I) | 20 Months
  Assessment of treatment effect with the change from baseline in Freiburg Visual Acuity (quantitative LogMAR score)

SECONDARY OUTCOMES:
Assessment of the effect of vMCO-I on functional vision outcomes | 20 Months
  Assessment of the treatment effect on the quality of Life with changes from baseline in activities of daily living using the National Eye Institute (NEI) Visual Function Questionnaire-25
Assessment of the durability of vMCO-I induced gene reporter expression | 20 Months
  Assessment of PK parameters including the Change in fundus fluorescence intensity of reporter (mCherry)

CONTACTS AND LOCATIONS:
Overall Officials: Samarendra Mohanty, Study Director — Nanoscope Therapeutics Inc.
Locations (1):
- JPM Rotary Club of Cuttack Eye Hospital and Research Institute, Cuttack, Odisha, India

IPD SHARING:
Plan to Share IPD: Yes
The results of the clinical trial will be made available when the study is completed and results are analyzed. The results will be published on this site and be available to conference presentations and publications.
Time Frame: Within a year from the long term monitoring data availability
Access Criteria: IPD sharing access will be subject to data transfer agreement. IPD generated as part of this clinical study may be subject to patient confidentiality.